CLINICAL TRIAL: NCT04248361
Title: A Randomized, Open-label, Multi-Center, Prospective Study to Assess the Clinical Utility of TEM-PCR™ Upper Respiratory Panel in Adult Patients 65 and Older Presenting With Symptoms of Acute Respiratory Illness
Brief Title: TEM-PCR™ Prospective Clinical Utility Study
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment due to COVID-19
Sponsor: Diatherix Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Diatherix-601
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-04

CONDITIONS: Upper Resp Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Multi-Center, Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TEM-PCR Diagnosis (Experimental): The TEM-PCR diagnostic technology will be used to assess for a source pathogen involved in the subject's acute respiratory illness. Results of the TEM-PCR URI Panel will be used by the physician to guide treatment decisions. If indicated, the investigator may also utilize rapid strep testing and rapid influenza testing for diagnosis. In the event a lower respiratory infection is suspected a chest x-ray or complete blood count (CBC) with differential may also be performed.
  Interventions: Diagnostic Test: TEM-PCR URI Panel
- SOC/Empiric Diagnosis (Active Comparator): The Standard of Care for upper respiratory infection may include, but is not limited to, rapid strep testing, rapid influenza testing, and sputum cultures. In the event a lower respiratory infection is suspected a chest x-ray or CBC with differential may be performed.
  Interventions: Other: SOC/Empiric Diagnosis

INTERVENTIONS:
Diagnostic Test: TEM-PCR URI Panel — Target Enriched Multiplex Polymerase Chain Reaction (TEM-PCR™) is a breakthrough molecular multiplex technology that allows rapid DNA/RNA identification of multiple pathogens (i.e., bacteria and viruses) in a single sample, typically within one day of specimen receipt.
  Arms: TEM-PCR Diagnosis
Other: SOC/Empiric Diagnosis — The SOC for upper respiratory infection may include, but is not limited to, rapid strep testing, rapid influenza testing, and sputum cultures. In the event a lower respiratory infection is suspected a chest x-ray or CBC with differential may be performed.
  Arms: SOC/Empiric Diagnosis

SUMMARY:
This is a randomized, open-label, multi-center, prospective study to assess the clinical utility of the TEM-PCR Upper Respiratory Infection (URI) Panel in adult subjects age 65 and older presenting to the primary care clinic with symptoms of acute respiratory illness.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, prospective study to assess the clinical utility of the TEM-PCR URI Panel in adult subjects age 65 and older presenting to the primary care clinic with symptoms of acute respiratory illness. The study will enroll 314 subjects with <10% of subjects having chronic conditions that may affect the lungs (i.e., CHF, COPD, and neoplastic disease of the lungs).

Subjects recruited from the general patient population visiting identified primary care clinic sites will be recruited and randomized to either TEM-PCR or Standard of Care (SOC)/empiric diagnosis for determination of respiratory pathogen(s). The treating physician will use the results of either the TEM-PCR panel or the SOC/empiric diagnosis to guide treatment decisions. Sputum sample (or nasopharyngeal swab if sputum sample cannot be collected) results obtained from the TEM-PCR diagnosis will be available in approximately one business day of sample collection. Sputum sample (or nasopharyngeal swab if sputum sample cannot be collected) results obtained from the SOC/empiric diagnosis will be available in approximately 3-5 business days of sample collection. The Investigator may call the subject upon receipt of sputum sample results if the results indicate that a change in therapy is necessary. All changes in the prescribed treatment plan will be documented in the subject's source documents. Subjects will record all therapy used for the treatment of respiratory illness and adverse events from Day 1 through Day 30 in a patient diary.

A final in-clinic visit will be conducted on Day 30 (± 5 days) following the Day 1 clinic visit to assess for outcomes (i.e., antibiotic treatment and duration/completion, use of antivirals and duration/completion, rate of clinic revisit or hospital admission and subsequent length of stay, mortality rate, use of steroids and/or antipyretics, use of OTC symptomatic treatments, and use of supportive therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent for the trial;
2. Age 65 years or older;
3. In the opinion of the investigator, subject has the cognitive ability to provide accurate information to study site personnel and to follow instructions, or subject has a caregiver who can provide accurate information and ensure subject's compliance with instructions;
4. Presentation with at least two of the following symptoms of acute respiratory illness:

   1. nasal congestion
   2. chest congestion
   3. shortness of breath
   4. cough
   5. body ache
   6. fever (≥100.4 ºF)

Exclusion Criteria:

1. Subject is currently taking antibiotics or has taken antibiotics within the previous 30 days.
2. Subject is currently taking antivirals or has taken antivirals within the previous 30 days.
3. Subject has been hospitalized within the previous 30 days.
4. Severity of illness (according to the Investigator) requires immediate hospitalization or referral to specialty care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with revisit to a healthcare facility | 30 days
  The rate of revisit to a healthcare facility (i.e., revisit to primary care, urgent care, or hospital ER) for the same reason (respiratory infection) as the initial visit between subjects assigned to SOC/empiric diagnosis and TEM-PCR diagnosis as well as in a subset of subjects with bacterial superinfection

SECONDARY OUTCOMES:
Proportion of subjects prescribed antibiotics on Day 1 for respiratory infection | 30 days
Proportion of subjects prescribed or continuing antibiotics for respiratory infection on the day of pathogen diagnosis | 30 days
Total number of days of antibiotic use for respiratory infection during the follow-up period | 30 days
Appropriateness of initial antibiotic selection for respiratory infection | 30 days
  Appropriateness will be determined by the investigator based upon pathogen sensitivity to the initial antibiotic selection as determined by sputum culture results.
Proportion of subjects prescribed antivirals (i.e., oseltamivir, zanamivir, etc.) for respiratory infection on Day 1 | 30 days
Proportion of subjects prescribed or continuing antivirals for respiratory infection on the day of pathogen diagnosis | 30 days
Total number of days of antiviral use for respiratory infection during the follow-up period | 30 days
Appropriateness of initial antiviral selection for respiratory infection | 30 days
  Appropriateness will be determined by the investigator based upon pathogen sensitivity to the initial antiviral selection as determined by sputum culture results.
Hospital admission for respiratory infection | 30 days
  The subject will be assessed as to whether or not they were admitted to a hospital during the time from the initial clinic visit until the final Day 30 clinic visit.
Mortality from any cause within 30 days of Clinic visit | 30days
Clearance of respiratory infection at 30 days | 30 days
  The investigator will assess the patient via a directed physical exam to assess whether the patient's respiratory infection has resolved. This assessment will be conducted at the Day 30 visit.
Use (or increase in use) of steroids and/or antipyretics (acetaminophen/NSAIDs) for the treatment of respiratory illness | 30 days
Use of OTC symptomatic treatment (i.e., antitussives, decongestants, and antihistamines) for the treatment of respiratory illness | 30 days
Use of supportive care (i.e., mechanical ventilation, addition of oxygen therapy or increase in oxygen use) | 30 days
Length of hospital stay for respiratory infection | 30 days
  If a subject is admitted to the hospital for respiratory infection at any point from the initial clinic visit until the final Day 30 clinic visit, the length of the admission (in days) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Hassoun, MD, Principal Investigator — Alabama Infectious Disease Center
Locations (4):
- United States (4):
  - Twilight Medical Center, Athens, Alabama
  - Valley Internal Medicine, Athens, Alabama
  - Blankenship Family Medicine, Huntsville, Alabama
  - Comprehensive Primary Care and Urgent Care of Alabama, Huntsville, Alabama

IPD SHARING:
Plan to Share IPD: No